CLINICAL TRIAL: NCT04411251
Title: Integrative Oncology - Evaluation of a Oncology Day Care Unit Programme With Two Different Focuses
Brief Title: Evaluation of a Oncology Day Care Unit Programme With Two Different Focuses
Acronym: TK-Onko
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TK-Onko
Record Dates: First submitted 2020-05-25; First posted 2020-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Cancer
Keywords: Nature; Mind-Body Therapies; Mindfulness; Yoga; Meditation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outdoor (Experimental): Nature-centered therapy in a near-natural area
  Interventions: Behavioral: Nature-near integrative day care unit programme
- Indoor (Active Comparator): Conventional therapy in rooms mainly in a hospital building
  Interventions: Behavioral: Conventional integrative day care unit programme

INTERVENTIONS:
Behavioral: Nature-near integrative day care unit programme — Interventions based on the Mind Body Medicine in Integrative and Complementary Medicine (MICOM) programme
  Arms: Outdoor
Behavioral: Conventional integrative day care unit programme — Interventions based on the Mind Body Medicine in Integrative and Complementary Medicine (MICOM) programme
  Arms: Indoor

SUMMARY:
The aim of this study is to investigate the effects of a nature-centred integrative oncology day care unit programme ("outdoor concept") compared with an already established integrative oncology day care unit programme ("indoor concept").

ELIGIBILITY:
Inclusion Criteria:

- cancer diagnosis

Exclusion Criteria:

* cognitive impairment that would interfere with questionnaire replies or the intervention
* pregnancy or lactation
* known serious mental illness
* participation in another study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - General (FACT-G) | Change from date of inclusion (baseline) at 12 weeks and at 24 weeks
  Assessing full scale, range 0-108, higher score meaning a better outcome

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-40, higher score meaning a better outcome
Functional Assessment of Cancer Therapy: Fatigue (FACT-F) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-52, higher score meaning a better outcome
WHO-Five Well-Being Index (WHO-5) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-25, higher score meaning a better outcome
Perceived Benefits of Nature Questionnaire (PBNQ) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  mean score of the 11 items, range 1-7, lower score meaning a better outcome
Perceived Stress Scale (PSS-10) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-40, lower score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-42, lower score meaning a better outcome
Flourishing Scale (FS-D) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 8-56, higher score meaning a better outcome
Freiburg Mindfulness Inventory (FMI) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-56, higher score meaning a better outcome
Insomnia Severity Index (ISI) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-28, lower score meaning a better outcome
Self-Efficacy Scale - Short Form (ASKU) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  mean score of the 3 items, range 1-5
Self-Compassion Scale (SCS-D) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  mean score of 12 items, range 1-5, higher score meaning a better outcome
Behavioral questions: alcohol consumption | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Number of alcoholic beverages on average per week in the last month
Behavioral questions: relaxation | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Relaxation behavior on average per week in the last month in minutes
Behavioral questions: cigarettes | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Number of cigarettes on average per week in the last month in minutes
Sociodemographic Measurements | Date of inclusion (baseline)
  Age, gender, education level, household income, employment status, marital status, complete family history, current and previous diseases and co-morbidities, current medication intake
Body weight | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  kg
Expectation questions | Date of inclusion (baseline)
  For intervention 1 and intervention 2 on a 5-point likert scale from 1 (nothing at all) to 5 (very strong)
Behavioral questions: sport | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Sports behavior on average per week in the last month in minutes

OTHER OUTCOMES:
Qualitative interviews | 12 weeks and 24 weeks after inclusion
  Qualitative assessment will be carried out in qualitative interviews in 20 patients participating in the study. The interviews will be recorded, transcribed and analyzed with qualitative content analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes